CLINICAL TRIAL: NCT01565850
Title: A Phase 2, Randomized, Double-Blinded Study of the Safety and Efficacy of Darunavir/Cobicistat/Emtricitabine/GS-7340 Single Tablet Regimen Versus Cobicistat-boosted Darunavir Plus Emtricitabine/Tenofovir Disoproxil Fumarate Fixed Dose Combination in HIV-1 Infected, Antiretroviral Treatment Naive Adults
Brief Title: D/C/F/TAF Versus COBI-boosted DRV Plus FTC/TDF in HIV-1 Infected, Antiretroviral Treatment Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-299-0102
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment-Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Darunavir; Cobicistat; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D/C/F/TAF (Experimental): D/C/F/TAF FDC tablet plus DRV placebo plus COBI placebo plus FTC/TDF placebo
  Interventions: Drug: D/C/F/TAF; Drug: DRV Placebo; Drug: COBI Placebo; Drug: FTC/TDF Placebo
- DRV+COBI+FTC/TDF (Active Comparator): DRV tablet plus COBI tablet plus FTC/TDF 200/300 mg FDC tablet plus D/C/F/TAF placebo
  Interventions: Drug: DRV; Drug: COBI; Drug: FTC/TDF; Drug: D/C/F/TAF Placebo

INTERVENTIONS:
Drug: D/C/F/TAF — DRV 800 mg/COBI 150 mg/FTC 200 mg/TAF 10 mg FDC tablet administered orally once daily
  Arms: D/C/F/TAF
Drug: DRV — DRV 800 mg (2 × 400 mg tablets) administered orally once daily
  Other Names: Prezista®
  Arms: DRV+COBI+FTC/TDF
Drug: COBI — COBI 150 mg tablet administered orally once daily
  Other Names: Tybost®; GS-9350
  Arms: DRV+COBI+FTC/TDF
Drug: FTC/TDF — FTC 200 mg/TDF 300 mg FDC tablet administered orally once daily
  Other Names: Truvada®
  Arms: DRV+COBI+FTC/TDF
Drug: D/C/F/TAF Placebo — D/C/F/TAF placebo tablet administered orally once daily
  Arms: DRV+COBI+FTC/TDF
Drug: DRV Placebo — DRV placebo tablet administered orally once daily
  Arms: D/C/F/TAF
Drug: COBI Placebo — COBI placebo tablet administered orally once daily
  Arms: D/C/F/TAF
Drug: FTC/TDF Placebo — FTC/TDF placebo tablet administered orally once daily
  Arms: D/C/F/TAF

SUMMARY:
This study is to evaluate the safety and efficacy darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) fixed dose combination (FDC) tablet versus darunavir (DRV)+cobicistat (COBI)+emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) in HIV-1 infected, antiretroviral treatment-naive adults as determined by the achievement of HIV-1 RNA < 50 copies/mL at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) males or non-pregnant females
* Ability to understand and sign a written informed consent form
* General medical condition which does not interfere with the assessments and the completion of the trial
* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL
* CD4+ cell count > 50 cells/µL
* Treatment-naive: No prior use of any approved or experimental anti-HIV drug for any length of time
* Screening genotype report must show sensitivity to DRV, TDF and FTC
* Normal ECG
* Adequate renal function: Estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft Gault formula
* Hepatic transaminases ≤ 2.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL
* Serum amylase ≤ 5 x ULN
* Adequate hematologic function
* Normal thyroid-stimulating hormone (TSH)
* Females of childbearing potential must have a negative serum pregnancy test
* Females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 30 days following the last dose of study drugs
* Female subjects who are postmenopausal must have documentation of cessation of menses for ≥ 12 months and hormonal failure
* Female subjects who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level test
* Male subjects must agree to utilize a highly effective method of contraception during heterosexual intercourse throughout the study period and for 90 days following discontinuation of investigational medicinal product

Exclusion Criteria:

* A new AIDS defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen positive
* Hepatitis C antibody positive
* Proven acute hepatitis in the 30 days prior to study entry
* Have a history or experiencing decompensated cirrhosis
* Current alcohol or substance use that potentially interferes with study compliance
* Any other clinical condition or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing requirements
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Female subjects who utilize non-estrogen hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Have an implanted defibrillator or pacemaker
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Baseline
* Participation in any other clinical trial without prior approval is prohibited while participating in this trial
* Receiving ongoing therapy with any of the disallowed medications, including drugs not to be used with darunavir and cobicistat
* Note: darunavir is a sulfonamide. Participants who previously experienced a sulfonamide allergy will be allowed to enter the trial. To date, no potential for cross sensitivity between drugs in the sulfonamide class and darunavir has been identified in patients participating in Phase 2 and Phase 3 trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moupali Das, MD, MPH, Study Director — Gilead Sciences
Locations (44):
- United States (43):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - AHF Research Center, Beverly Hills, California
  - Kaiser Permanente, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alta Bates Summit Medical Center, East Bay AIDS Center, Oakland, California
  - Stanford University, Palo Alto, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Kasier Permanente Medical Center, San Francisco, California
  - TPMG--Clinical Trials Unit, San Francisco, California
  - Apex Research, Denver, Colorado
  - Denver Infectious Disease Consultants, PLLC, Denver, Colorado
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Gary J. Richmond,M.D.,P.A., Fort Lauderdale, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ValuhealthMD, LLC, Orlando, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University Mercer Medicine, Macon, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Community Research Initiative (CRI), Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research Inc, St Louis, Missouri
  - North Shore University Hospital / Division of Infectious Diseases, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - ID Consultants, P.A., Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of South Carolina School of Medicine Division of Infectious Disease, Columbia, South Carolina
  - Southwest Infectious Disease Clinical Research Inc, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot, MD., PA, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - CARE-ID, Annandale, Virginia
  - Peter Shalit, M.D., Seattle, Washington
- Clinical Research Puerto Rico, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States (including Puerto Rico). The first participant was screened on 16 April 2012. The last study visit occurred on 19 February 2014.
Pre-assignment Details: 232 participants were screened.
Groups:
- D/C/F/TAF: Darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) (800/150/200/10 mg) fixed-dose combination (FDC) tablet plus darunavir (DRV) placebo plus cobicistat (COBI) placebo plus emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) placebo once daily
- DRV+COBI+FTC/TDF: DRV 800 mg tablet plus COBI 150 mg tablet plus FTC/TDF 200/300 mg FDC tablet plus D/C/F/TAF placebo once daily
Period: Overall Study
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Started | 103 | 50
Completed | 83 | 42
Not Completed | 20 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 12 | 4
Not completed — Investigator's Discretion | 2 | 1
Not completed — Participant noncompliance | 2 | 0
Not completed — Withdrew Consent | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Groups:
- D/C/F/TAF: D/C/F/TAF (800/150/200/10 mg) FDC tablet plus DRV placebo plus COBI placebo plus FTC/TDF placebo once daily
- Total: Total of all reporting groups
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF | Total
Number analyzed (Participants) | 103 | 50 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11.3) | 37 (10.9) | 35 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 95 | 47 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 9 | 32
  Not Hispanic or Latino | 80 | 41 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 62 | 30 | 92
  Black or African American | 36 | 17 | 53
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 103 | 50 | 153
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.70 (0.516) | 4.65 (0.514) | 4.68 (0.515)
HIV-1 RNA Category [Number; unit: participants]
  ≤ 100,000 copies/mL | 80 | 43 | 123
  > 100,000 to ≤ 400,000 copies/mL | 17 | 5 | 22
  > 400,000 copies/mL | 6 | 2 | 8
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 395 (169.3) | 464 (261.6) | 417 (205.7)
CD4 Cell Count Category [Number; unit: participants]
  < 50 cells/μL | 1 | 1 | 2
  50 to ≤ 199 cells/µL | 10 | 9 | 19
  200 to ≤ 349 cells/µL | 37 | 8 | 45
  351 to ≤ 499 cells/µL | 27 | 12 | 39
  ≥ 500 cells/μL | 28 | 20 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24
Description: The snapshot algorithm was used which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set: participant who were randomized;enrolled and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Number analyzed (Participants) | 103 | 50
percentage of participants | 74.8 | 74.0
Statistical Analysis 1: Comparison: D/C/F/TAF vs DRV+COBI+FTC/TDF; The null hypothesis was that the D/C/F/TAF group is at least 12% worse than the DRV+COBI+FTC/TDF group with respect to the percentage of participants achieving HIV-1 RNA < 50 copies/mL (response rate as defined by the snapshot analysis algorithm) at Week 24; the alternative hypothesis was that the response rate in the D/C/F/TAF group is less than 12% worse than that in the DRV+COBI +FTC/TDF group; Test type: Non-Inferiority or Equivalence — A total sample size of 150 HIV-1 infected participants, randomized in a 2:1 ratio to 2 groups, would achieve 56% power to evaluate noninferiority with respect to the response rate of HIV-1 RNA < 50 copies/mL at Week 24 if a response rate of 0.88 for both arms, a noninferiority margin of 0.12, and the significance level of the test at a one-sided 0.025 level were assumed; p = 0.64, Cochran-Mantel-Haenszel — The p-value for the superiority test comparing the percentages of virologic success was from the Cochran-Mantel-Haenszel test stratified by baseline HIV-1 RNA and race strata; Difference in proportions = 3.3, 95% CI 2-sided [-11.4 to 18.1] — The difference in percentages of virologic success and its 95% confidence interval (CI) were calculated based on baseline HIV-1 RNA and race stratum-adjusted Mantel-Haenszel proportion

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Number analyzed (Participants) | 103 | 50
percentage of participants | 76.7 | 84.0
Statistical Analysis 1: Comparison: D/C/F/TAF vs DRV+COBI+FTC/TDF; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the D/C/F/TAF group is at least 12% worse than the DRV+COBI+FTC/TDF group with respect to the percentage of participants achieving HIV-1 RNA < 50 copies/mL (response rate as defined by the snapshot analysis algorithm) at Week 48; the alternative hypothesis was that the response rate in the D/C/F/TAF group is less than 12% worse than that in the DRV+COBI +FTC/TDF group; p = 0.35, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in proportions = -6.2, 95% CI 2-sided [-19.9 to 7.4] — The difference in percentages of virologic success and its 95% CI were calculated based on baseline HIV-1 RNA and race stratum-adjusted Mantel-Haenszel proportion

3. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with Week 24 data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Number analyzed (Participants) | 92 | 48
log10 copies/mL | -3.20 (0.653) | -3.18 (0.416)
Statistical Analysis 1: Comparison: D/C/F/TAF vs DRV+COBI+FTC/TDF; Test type: Superiority or Other; p = 0.67, ANOVA — The p-value, difference in least squares mean (LSM), and its 95% CI were from ANOVA model with baseline HIV-1 RNA level (≤ 100,000 or > 100,000 copies/mL) and race (Black or non-Black) as fixed effects in the model; Difference in LSM = 0.04, 95% CI 2-sided [-0.14 to 0.21]

4. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with Week 48 data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Number analyzed (Participants) | 89 | 47
log10 copies/mL | -3.27 (0.668) | -3.26 (0.521)
Statistical Analysis 1: Comparison: D/C/F/TAF vs DRV+COBI+FTC/TDF; Test type: Superiority or Other; p = 0.50, ANOVA — The p-value, difference in LSM, and its 95% CI were from ANOVA model with baseline HIV-1 RNA level (≤ 100,000 or > 100,000 copies/mL) and race (Black or non-Black) as fixed effects in the model; Difference in LSM = 0.06, 95% CI 2-sided [-0.11 to 0.23]

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with Week 24 data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Number analyzed (Participants) | 91 | 48
cells/µL | 186 (137.9) | 139 (185.8)
Statistical Analysis 1: Comparison: D/C/F/TAF vs DRV+COBI+FTC/TDF; Test type: Superiority or Other; p = 0.11, ANOVA — [p-value comment as in outcome 4, analysis 1]; Difference in LSM = 45, 95% CI 2-sided [-10 to 101]

6. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with Week 48 data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Number analyzed (Participants) | 85 | 46
cells/µL | 231 (141.9) | 212 (151.5)
Statistical Analysis 1: Comparison: D/C/F/TAF vs DRV+COBI+FTC/TDF; Test type: Superiority or Other; p = 0.50, ANOVA — [p-value comment as in outcome 4, analysis 1]; Difference in LSM = 18, 95% CI 2-sided [-35 to 72]

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure: D/C/F/TAF group = 61.7 weeks; DRV+COBI+FTC/TDF group = 66.1 weeks) plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Arm/Group | D/C/F/TAF | DRV+COBI+FTC/TDF
Serious Adverse Events (participants affected / at risk) | 5/103 | 2/50
Other Adverse Events (participants affected / at risk) | 77/103 | 40/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF (N=103) | DRV+COBI+FTC/TDF (N=50)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D/C/F/TAF (N=103) | DRV+COBI+FTC/TDF (N=50)
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 22 | 13
Flatulence (Gastrointestinal disorders) | 5 | 6
Haemorrhoids (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 13 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5
Fatigue (General disorders) | 14 | 9
Pyrexia (General disorders) | 7 | 2
Bronchitis (Infections and infestations) | 9 | 2
Folliculitis (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 3
Pharyngitis (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 7 | 4
Tooth abscess (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 16 | 7
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 5
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Headache (Nervous system disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 12 | 4
Hypertension (Vascular disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years